CLINICAL TRIAL: NCT07243496
Title: Composite Restoration of Class II Cavities in Primary Molars With or Without Pulpotomy. Prospective 24 Month Clinical Trial.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lygidakis Dental Clinic (Other)
Responsible Party: Principal Investigator, Nikos Lygidakis, Dr, Lygidakis Dental Clinic
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1495
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Composite Restoration; Primary Tooth Pulpotomy
Keywords: class II cavity; primary tooth; pulpotomy
MeSH Terms: interventions — Pulpotomy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Class II composite restoration on primary teeth with pulpotomy (Active Comparator)
  Interventions: Procedure: Class II restoration after pulpotomy
- Class II composite restoration on primary teeth without pulpotomy (Active Comparator)
  Interventions: Procedure: Class II restoration without pulpotomy

INTERVENTIONS:
Procedure: Class II restoration after pulpotomy — The same dentist performs all restorations. All treatments are carried out using a rubber dam and the appropriate local anesthesia. After pulpotomy completion with a layer of MTA®, an intermediate layer of glass ionomer cement (Vitrebond Plus™) is placed before the final composite resin restoration. Class II resin restorations are performed after complete caries removal, placement of a partial matrix, etching with 37% phosphoric acid for 15 seconds, bonding with a 4th-generation adhesive agent (Prime n Bond NT, Dentsply™), and placement of composite resin (Filtek Universal™, 3M™).
  Arms: Class II composite restoration on primary teeth with pulpotomy
Procedure: Class II restoration without pulpotomy — The same dentist performs all restorations. All treatments are carried out using a rubber dam and the appropriate local anesthesia. Class II resin restorations are performed after complete caries removal, placement of a partial matrix, etching with 37% phosphoric acid for 15 seconds, bonding with a 4th-generation adhesive agent (Prime n Bond NT, Dentsply™), and placement of composite resin (Filtek Universal™, 3M™).
  Arms: Class II composite restoration on primary teeth without pulpotomy

SUMMARY:
After 24 months:

* Investigation of the success rate of Class II composite resin restorations in primary molars that have undergone pulpotomy.
* Comparison of Class II composite resin restorations in primary molars that have undergone pulpotomy with restorations of the same type in the same patient, in which no pulpotomy has been performed.

The null hypothesis of the study is that there is no statistically significant difference in the success of Class II resin restorations after their placement in primary molars, regardless of whether a pulpotomy has been performed or not.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged 3-9 years

  * At least one pulpotomy in a carious primary molar requiring a Class II resin restoration
  * At least one Class II cavity in a carious primary molar in the same patient that requires a resin restoration
  * The teeth to be restored must not present clinical signs of pulp necrosis, such as pathological mobility or abscess/fistula
  * Parents have signed an informed consent form
  * The young patients return for evaluation at 12 and 24 months
  * There is no exfoliation or extraction of the evaluated teeth before the 24-month period

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Modified USPHS criteria | Assessment is done at 12 and 24 months following placement of the composite restoration
  Modified USPHS criteria are variations of the original United States Public Health Service criteria used in dentistry to clinically evaluate restorations. They include the following criteria: marginal adaptation, retention, marginal discoloration, and secondary caries, with specific parameters and scoring scales adjusted for a particular study or material being evaluated. These modifications allow for a more precise assessment of dental restorations by tailoring the evaluation to specific clinical situations or restorative materials

CONTACTS AND LOCATIONS:
Locations (1):
- Lygidakis Dental Clinic, Athens, Greece

IPD SHARING:
Plan to Share IPD: No